CLINICAL TRIAL: NCT06355063
Title: Initial Safety and Performance of the CellFX® nsPFA™ Cardiac Surgery System for the Treatment of Atrial Fibrillation
Brief Title: CellFX® nsPFA™ Cardiac Surgery System to Treat Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-PCF-037; NCT06355063 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2024-04-01; First posted 2024-04-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Surgery; Ablation of Atrial Fibrillation; Clamp Study
Keywords: CellFX; nsPFA Cardiac Surgery System
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, single arm, non-randomized, feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CellFX nsPFA Treatment Arm (Experimental): Adult subjects who are clinically indicated for a concomitant cardiac surgical procedure will undergo left pulmonary vein, roof and floor ablations to form a left atrial posterior box using the CellFX® nsPFA™ Cardiac Surgery System.
  Interventions: Device: CellFX® nsPFA™ Cardiac Surgery System

INTERVENTIONS:
Device: CellFX® nsPFA™ Cardiac Surgery System — Adult patients presenting to the investigational center that are to undergo non-emergent concomitant cardiac surgical procedure(s), scheduled to be performed on cardiopulmonary bypass including open-heart surgery for one or more of the following: mitral valve repair or replacement, aortic valve repair or replacement, ascending aortic aneurysms, or coronary artery bypass procedures with history of documented atrial fibrillation within one year prior to enrollment will be evaluated for eligibility and participation in the study.

SUMMARY:
This feasibility study will be conducted to demonstrate the initial safety and effectiveness of the CellFX® nsPFA™ Cardiac Clamp in performing a box lesion around the 4 pulmonary veins as an isolated procedure or as a part of a more extensive surgical ablation set in conjunction with concomitant cardiac surgical procedure.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single arm, non-randomized, feasibility study. Adult subjects who are clinically indicated for a concomitant cardiac surgical procedure will undergo left pulmonary vein, roof and floor ablations to form a left atrial posterior box. All subjects will return to the hospital between 60-120 days post-surgical ablation procedure to undergo a cardiac electrophysiology study with electroanatomical mapping to assess electrical isolation of the pulmonary veins and left atrial posterior wall

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 and 85 years of age
* Subject is willing and capable of providing Informed Consent to undergo study procedures which includes surgical AF ablation and completing follow-up visits as specified in the clinical study protocol
* Subject has history of documented atrial fibrillation within one year prior to enrollment. Documentation may include ECG, transtelephonic monitor (TTM), holter monitor or telemetry strip
* Subject is scheduled to undergo non-emergent cardiac surgical procedure(s) to be performed on cardiopulmonary bypass including open-heart surgery for one or more of the following: Mitral valve repair or replacement, Aortic valve repair or replacement, Ascending aortic aneurysms, or Coronary artery bypass procedures
* Left ventricular ejection fraction ≥ 30% (determined by echocardiography or cardiac catheterization performed within 60 days of enrollment as documented in patient medical history)
* Subject has a life expectancy of at least 5 years

Exclusion Criteria:

* Subject has an implantable electronic medical device. (i.e., pacemaker, ICD or CRT) or left atrial appendage device
* Subject has a prosthetic heart valve
* Stand-alone AF without indication(s) for concomitant Coronary Artery Bypass Graft (CABG) and/or valve surgery
* Previous surgical Maze procedure
* Prior cardiac surgery (Redo)
* Wolff-Parkinson-White syndrome or other Supra-Ventricular arrhythmia, Atrioventricular (AV) nodal reentry
* Subjects requiring surgery other than CABG and/or cardiac valve surgery and/or atrial septal defect repair.
* Prior history of medical procedure involving instrumentation of the left atrium (e.g., previous ablation)
* Class IV New York Heart Association (NYHA) heart failure symptoms
* Prior history of cerebrovascular accident or TIA within 6 months or at any time if there is residual neurological deficit
* Documented ST-segment elevation Myocardial Infarction (MI) within the 6 weeks prior to study enrollment
* Need for emergent cardiac surgery (i.e., cardiogenic shock)
* Known carotid artery stenosis greater than 80%
* Current diagnosis of active systemic infection
* Severe peripheral arterial occlusive disease defined as claudication with minimal exertion
* Renal failure requiring dialysis or hepatic failure
* A known drug and/or alcohol addiction
* Mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study
* Pregnancy or desire to get pregnant within 12-months of the study treatment
* Preoperative need for an intra-aortic balloon pump or intravenous inotropes
* Subjects who have been treated with thoracic radiation
* Subjects in current chemotherapy
* Subjects on long term treatment with oral or injected steroids (not including intermittent use of inhaled steroids for respiratory diseases)
* Subjects with known hypertrophic obstructive cardiomyopathy
* Subjects with known cold agglutinin
* History of abnormal bleeding and/or clotting disorder
* Contraindication to anticoagulation (i.e., Heparin, Dabigatran, Apixaban, Vitamin K Antagonists such as warfarin)
* Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
* Body mass index > 40 kg/m2
* Use of any other investigational drug, therapy, or device within 30 days prior to enrollment or concurrent participation in another research study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of acute major adverse events (MAEs) | Within 30 days post-ablation procedure
  Acute major adverse events (MAEs) include, cardiac death, stroke, myocardial infarction, transient ischemic attack, or excessive bleeding.
Number of Participants with acute electrical isolation of the bilateral pulmonary veins and left atrial box | Within 24 hours post-ablation procedure
  The ablation procedure includes pulmonary vein isolation and a series of ablation lines to create a "box lesion" on the posterior left atrial free wall. At the conclusion of both the primary and concomitant procedures, exit and/or entrance block will be performed to confirm complete isolation of the pulmonary veins and the left atrial posterior wall.

SECONDARY OUTCOMES:
Proportion of Participants with one or more SAEs | Up to 12-months post-procedure
  Long-term safety endpoint for the incidence of treatment-emergent adverse events [Safety and Tolerability] for subjects having one or more SAEs at each follow-up interval.
Number of Participants with Long-Term Technical Success | 60-120 days following the index procedure
  Long-term Technical Success of the Pulse Biosciences CellFX® nsPFA™ Cardiac Surgery System is defined as participants having confirmation of electrical isolation of the bilateral pulmonary veins and left atrial box by cardiac electroanatomical mapping 2-6 months post-ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rich Nuccitelli, PhD, Study Director — Pulse Biosciences, Inc.
Locations (6):
- Medical University of Vienna, Vienna, Austria
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Catharina Hospital, Eindhoven
  - Maastricht University Medical Center+ (MUMC+), Maastricht
  - St. Antonius Hospital, Nieuwegein
- State Medical Institute of the Ministry of Interior Affairs and Administration, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No